CLINICAL TRIAL: NCT03711331
Title: Impact of a Strategy Based on the Unyvero® Testing System on Appropriate and Targeted Antimicrobial Treatment in Patients With Suspected VAP or HAP Requiring Mechanical Ventilation: a Randomized Controlled Unblinded Trial
Brief Title: Impact of a Strategy Based on Bacterial DNA Detection to Optimize Antibiotics in Patients With Hospital-acquired Pneumonia
Acronym: VAPERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Curetis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017_37; 2018-A00149-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia, Ventilator-Associated; Pneumonia, Bacterial
Keywords: Ventilator-associated pneumonia; Hospital-acquired pneumonia; Antimicrobial therapy; Ventilator-associated pneumonia Hospital-acquired pneumonia Antimicrobial therapy Polymerase chain reaction Antibiotics stewardship; Polymerase chain reaction; Antibiotics stewardship
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia, Bacterial; Healthcare-Associated Pneumonia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FilmArray® Pneumonia panel plus strategy (Experimental): patients benefiting from the new strategy based on the system Unyvero ®
  Interventions: Other: FilmArray® Pneumonia panel plus
- Standard care (Sham Comparator): patients benefiting from usual standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Other: FilmArray® Pneumonia panel plus — Early adjustment of antimicrobial therapy according to the results of the Unyvero® testing for patients suspected with VAP or HAP requiring MV.
  Arms: FilmArray® Pneumonia panel plus strategy
Other: Standard care — Standard care, with broad-spectrum antimicrobial therapy unchanged until reception of traditional microbiology results
  Arms: Standard care

SUMMARY:
VAPERO is a randomized, unblinded, controlled study to measure the impact of a strategy based on the Unyvero® multiplex PCR test on the adjustment of antimicrobial therapy in patients suspected with ventilator-associated or hospital-acquired pneumonia (VAP/HAP) requiring mechanical ventilation. The gold-standard microbiological diagnostic method for pneumonia in the ICU is still culture-based identification and antimicrobial susceptibility testing (AST) despite being more than a hundred years old, with results turnaround time spanning over several days, exposing patients to potentially inappropriate broad-spectrum antimicrobial therapy. The investigators aim to measure the impact of the Unyvero® testing strategy to improve the percentage of patients with VAP or HAP receiving early targeted antimicrobial therapy compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized in the ICU
* suspected with VAP or HAP requiring MV

Exclusion Criteria:

* Severe immunodeficiency
* Moribund patients (SAPS II > 90)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with targeted antibiotics regimen 24 hours after starting antimicrobial therapy in the experimental group compared to control group | 24 hours after the initiation of empiric antimicrobial therapy

SECONDARY OUTCOMES:
Percentage of patients receiving appropriate antimicrobial therapy 24 hours after antibiotics initiation | 24 hours after antibiotics start Daily until 7 days after antibiotics start 14 days after antibiotics start 28 days after antibiotics start
Amount of days alive and free from mechanical ventilation at day 28 after antibiotics initiation. | 24 hours after antibiotics start Daily until 7 days after antibiotics start 14 days after antibiotics start 28 days after antibiotics start
Length of stay in Intensive Care Unit | 24 hours after antibiotics start Daily until 7 days after antibiotics start 14 days after antibiotics start 28 days after antibiotics start
Number of Patient Deaths | at 28 days after antibiotics start
  number of patient deaths after antibiotics start
number of patient deaths in ICU | 24 hours after antibiotics start Daily until 7 days after antibiotics start 14 days after antibiotics start 28 days after antibiotics start

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU Lille, Lille, France

REFERENCES:
- [Background] Kerneis S, Visseaux B, Armand-Lefevre L, Timsit JF. Molecular diagnostic methods for pneumonia: how can they be applied in practice? Curr Opin Infect Dis. 2021 Apr 1;34(2):118-125. doi: 10.1097/QCO.0000000000000713. PMID 33395094